CLINICAL TRIAL: NCT01158482
Title: FILTER - Filter Initial & Long Term Evaluation After Placement and Retrieval (Including Laser-Assisted Retrieval) Prospective Registry
Brief Title: Filter Initial & Long Term Evaluation After Placement and Retrieval Registry
Acronym: FILTER
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, William Kuo, M.D., Stanford University
Other Study IDs: SU-06252010-6416; 19051 - eProtocol; FILTER REGISTRY (Other: STANFORD)
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IVC Filter Placement or Removal: Patients undergoing IVC filter placement and/or IVC filter removal at Stanford Medical Center.
  Interventions: Procedure: IVC Filter Placement or Retrieval

INTERVENTIONS:
Procedure: IVC Filter Placement or Retrieval — An IVC Filter will be placed or removed using endovascular techniques.

SUMMARY:
A prospective data registry for all patients who undergo IVC (Inferior Vena Cava) filter placement or retrieval at Stanford. Potential enrollees will already be undergoing the procedure. If patients are willing, they will be prospectively enrolled prior to the procedure. As part of the study, chart and clinical data reviews will be used to track patient progress and response to the treatment.

DETAILED DESCRIPTION:
Patient clinical data will be used in a clinical registry. Before a patient is to undergo their initial procedure for filter placement/retrieval, we will approach them for consent to participate in the study. If patients consent, we will follow clinical data from the procedure, and perform prospective follow-up over time to track clinical response and effects of the placement or removal procedure.

Various real-world protocols involving advanced filter removal (including laser-assisted filter removal) will be investigated by conducting registry-based clinical trials.

Participants will only be enrolled if they will be undergoing an IVC (Inferior Vena Cava) filter placement/retrieval procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participants are adults, 18 years old or older
* Participants will be undergoing a procedure to have an IVC filter placed or removed

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No specific criteria. Anyone who will be undergoing IVC Filter Placement/Retrieval will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2010-06; Primary Completion 2027-06 (Estimated); Study Completion 2030-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: William T Kuo MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Kuo WT, Doshi AA, Ponting JM, Rosenberg JK, Liang T, Hofmann LV. Laser-Assisted Removal of Embedded Vena Cava Filters: A First-In-Human Escalation Trial in 500 Patients Refractory to High-Force Retrieval. J Am Heart Assoc. 2020 Dec 15;9(24):e017916. doi: 10.1161/JAHA.119.017916. Epub 2020 Nov 30. PMID 33252283
- [Derived] Sheu AY, Hoang NS, Kesselman AJ, Liang T, Rosenberg JK, Kuo WT. Prophylactic IVC filter placement in bariatric surgery patients: results from a prospective filter registry. CVIR Endovasc. 2018;1(1):13. doi: 10.1186/s42155-018-0021-5. Epub 2018 Nov 15. PMID 30652145
- [Derived] Kuo WT, Odegaard JI, Rosenberg JK, Hofmann LV. Laser-Assisted Removal of Embedded Vena Cava Filters: A 5-Year First-in-Human Study. Chest. 2017 Feb;151(2):417-424. doi: 10.1016/j.chest.2016.09.029. Epub 2016 Oct 8. PMID 27729265
- [Derived] Kuo WT, Odegaard JI, Rosenberg JK, Hofmann LV. Excimer laser-assisted removal of embedded inferior vena cava filters: a single-center prospective study. Circ Cardiovasc Interv. 2013 Oct 1;6(5):560-6. doi: 10.1161/CIRCINTERVENTIONS.113.000665. Epub 2013 Sep 24. PMID 24065445